CLINICAL TRIAL: NCT04324580
Title: Postoperative Immobilization and Physical Therapy Following Volar Locked Plating for Distal Radius Fractures: Are They Necessary?
Brief Title: Postoperative Immobilization and Physical Therapy Following Volar Locked Plating for Distal Radius Fractures
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: NYU Langone Health (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 19-01584
Record Dates: First submitted 2020-03-05; First posted 2020-03-27 (Actual); Last update posted 2025-04-11 (Actual); Status verified 2025-04

CONDITIONS: Distal Radius Fracture
MeSH Terms: conditions — Wrist Fractures | interventions — Splints

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Delayed mobilization/Formal physical therapy group (Active Comparator): Participants will be placed into a volar-based plaster splint post-operatively. Participants will be asked to keep non-weight bearing (on the operated wrist) but no restrictions for range of motion, keeping the dressing in place until first post-operative visit at 2 weeks. After that, participants will be placed into a custom thermoplastic splint by a therapist. This will be worn for 5 weeks. Supervised physical therapy will be prescribed 1- 2 times per week for a total of 8 weeks along with a home exercise program. Active range of motion and strengthening exercises will be performed at home twice daily for 20 minutes for a total of 8 weeks. The splint will be removed only for formal and home physical therapy and hygiene.
  Interventions: Other: Splint; Behavioral: Formal Physical Therapy
- Immediate mobilization/self guided physical therapy group (Active Comparator): Participants will be placed into a soft dressing after surgery. Participants will be asked to keep non-weight bearing (on the operated wrist) but no restrictions for range of motion, keeping the dressing in place until first post-operative visit at 2 weeks. This group will be given a pamphlet with detailed instructions and demonstrations in home exercises. Active range of motion and strengthening exercises will be performed twice daily for 20 minutes for a total of 8 weeks.
  Interventions: Behavioral: Self directed physical therapy; Other: Soft dressing (No Splint)

INTERVENTIONS:
Other: Splint — Participants will have their open reduction internal fixation of distal radius fractures treated with volar locked plating. for 2 weeks. Which will be replaced by a custom thermoplastic splint for 5 weeks.
  Arms: Delayed mobilization/Formal physical therapy group
Behavioral: Formal Physical Therapy — Participants will also receive a prescription for formal physical therapy. Supervised physical therapy will be prescribed 1- 2 times per week for a total of 8 weeks along with a home exercise program. Active range of motion and strengthening exercises will be performed at home twice daily for 20 minutes for a total of 8 weeks.
  Arms: Delayed mobilization/Formal physical therapy group
Behavioral: Self directed physical therapy — Participants will be given a pamphlet with detailed instructions and demonstrations in home exercises. Active range of motion and strengthening exercises will be performed twice daily for 20 minutes for a total of 8 weeks.
  Arms: Immediate mobilization/self guided physical therapy group
Other: Soft dressing (No Splint) — Participants will have their open reduction internal fixation of distal radius fractures placed in a soft dressing which will be kept in place for 2 weeks.
  Arms: Immediate mobilization/self guided physical therapy group

SUMMARY:
The purpose of this study is to see if splinting and formal physical therapy are necessary following surgical fixation (open reduction internal fixation) of distal radius fractures (broken wrist). Currently there is no consensus for post-operative protocol following fixation of distal radius fractures. The decision to splint (late mobilization) and prescribe formal physical therapy vs. not to splint (early mobilization) and use self-guided physical therapy is based on surgeon or institutional preference. The goal of this study is to determine if early mobilization leads to improved outcomes and decreased costs without increasing pain or the loss of hardware fixation.

DETAILED DESCRIPTION:
188 patients treated for distal radius fractures with open reduction internal fixation using volar locked plating will be split into two study groups: a group that is immobilized in a splint post operatively and given formal physical therapy and a group that does not receive either of these post operative interventions. The primary outcome will be loss of fixation. Secondary outcomes will include pain, cost, Quick Dash, range of motion, and grip strength. Data will be recorded at the pre-operative visit, as well as at post-operative visits at 2 weeks, 6 weeks, 3 months and 6 months.

ELIGIBILITY:
Inclusion Criteria:

* Isolated displaced distal radius fractures, +/- ulnar styloid fracture, treated with volar locked plating and screws.

  1. > 10 degrees of dorsal tilt
  2. Volar displacement (Volar Barton's type fracture)
  3. Shortening > 3 mm
  4. Intra-articular displacement or step off > 2mm.

     Exclusion Criteria:
* Ipsilateral upper limb concomitant fracture
* Fracture fixation other than volar locked plating and screws
* Dislocation or neurologic injury
* Gustilo-Anderson grade III open fractures

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 230 (Actual)
Dates: Start 2020-06-18 (Actual); Primary Completion 2025-08-01 (Estimated); Study Completion 2025-08-01 (Estimated)

PRIMARY OUTCOMES:
Percentage of Loss of fixation | 2 weeks, 4 weeks, 12 weeks, 24 weeks
  The loss of fixation will be measured by the change in radiologic outcomes (in degrees) from 2-week post-operative visit to follow-up visits.

SECONDARY OUTCOMES:
Change in Patient comfort/pain (VAS) | Day of Surgery, 2 weeks, 4 weeks, 12 weeks, 24 weeks
  This will be measured by the Visual Analogue Scale (VAS) which measures pain using a 10 point scale. On a scale of 1-10 where following pain scale is: no pain (0), mild pain(1-3), moderate pain (4-6), and severe pain (7-10).
Change in wrist range mobility | 2 weeks, 4 weeks, 12 weeks, 24 weeks
  Range of motion will be measured using goniometers.
Change in wrist range mobility using DASH | 2 weeks, 4 weeks, 12 weeks, 24 weeks
  This is measured using the Disabilities of the Arm, Shoulder and Hand (DASH) questionnaire is a self-report questionnaire that patients can rate difficulty and interference with daily life on a 5 point Likert scale.
Change in Grip strength | 2 weeks, 4 weeks, 12 weeks, 24 weeks
  Physical examinations through the study will record the grip strength (kgs)

CONTACTS AND LOCATIONS:
Overall Officials: Jadie De Tolla, MD, Principal Investigator — NYU Langone Health
Locations (1):
- NYU Langone, New York, New York, United States

IPD SHARING:
Plan to Share IPD: Yes
Individual participant data that underlie the results reported in this article, after deidentification (text, tables, figures, and appendices).
Supporting Information: Study Protocol, SAP
Time Frame: Beginning 9 months and ending 36 months following article publication or as required by a condition of awards and agreements supporting the research.
Access Criteria: The investigator who proposed to use the data. Upon reasonable request. Requests should be directed to jadie.detolla@nyulangone.org To gain access, data requestors will need to sign a data access agreement.